CLINICAL TRIAL: NCT05329259
Title: A PHASE 4, OPEN-LABEL, SINGLE-ARM, MULTICENTER STUDY TO DESCRIBE THE SAFETY OF 13-VALENT PNEUMOCOCCAL CONJUGATE VACCINE IN ADULTS 18 TO 49 YEARS OF AGE IN INDIA
Brief Title: A Study to Describe the Safety of a Vaccine (Called 13vPnC) in Healthy People 18 to 49 Years of Age in India
Status: Completed | Phase: Phase 4 | Type: Interventional
Sponsor: Pfizer (Industry)
Responsible Party: Sponsor
Allocation: Not Applicable | Model: Single Group | Masking: None | Purpose: Prevention
Other Study IDs: B1851214
Record Dates: First submitted 2022-04-07; First posted 2022-04-14 (Actual); Results first posted 2024-04-26 (Actual); Last update posted 2024-04-26 (Actual); Status verified 2023-11

CONDITIONS: Pneumococcal Disease
MeSH Terms: conditions — Pneumococcal Infections

STUDY DESIGN:
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (1):
- 13-valent pneumococcal conjugate vaccine (Experimental): Pneumococcal conjugate vaccine (13vPnC)
  Interventions: Biological: 13-valent pneumococcal conjugate vaccine

INTERVENTIONS:
Biological: 13-valent pneumococcal conjugate vaccine — One dose of 13vPnC (0.5mL) will be administered intramuscularly.

SUMMARY:
* The purpose of this study is to describe the safety of the study vaccine (called 13vPnC) in people who are 18-49 years of age in India.
* This study is seeking participants who are generally healthy adults ≥18 and <50 years of age, with no prior history of pneumococcal vaccination.
* Participants will take part in the study for approximately one month which includes two visits to the study clinic.
* Participants will receive a single dose of study vaccine (13vPnC) into the arm at visit 1 and will come to study site for a follow-up visit after about a month.

ELIGIBILITY:
Inclusion Criteria:

* Generally healthy participants between the ages of ≥18 and <50 years at the time of consent.
* Participants who are determined by medical history, physical examination (if required), and clinical judgment of the investigator to be eligible for inclusion in the study.

Exclusion Criteria:

* History of severe adverse reaction associated with a vaccine and/or severe allergic reaction (eg, anaphylaxis) to any component of 13vPnC, or to any other diphtheria toxoid-containing vaccine.
* Congenital, functional, or surgical asplenia.
* Other medical or psychiatric condition including recent (within the past year) or active suicidal ideation/behavior or laboratory abnormality that may increase the risk of study participation or, in the investigator's judgment, make the participant inappropriate for the study.
* Previous vaccination with any pneumococcal vaccine, or planned receipt of any pneumococcal vaccine through study participation.

Ages: 18 Years to 49 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Adult
Enrollment: 200 (Actual)
Dates: Start 2022-10-06 (Actual); Primary Completion 2022-11-30 (Actual); Study Completion 2022-11-30 (Actual)

CONTACTS AND LOCATIONS:
Overall Officials: Pfizer CT.gov Call Center, Study Director — Pfizer
Locations (5):
- India (5):
  - Nirmal Hospital Pvt Ltd., Surat, Gujarat
  - BGS Global Institute of Medical Sciences (BGSGIMS), Bangalore, Karnataka
  - Jawahar Lal Nehru Medical College, Ajmer, Rajasthan
  - Calcutta School of Tropical Medicine, Kolkata, West Bengal
  - Aakash Healthcare Private Limited, Delhi

IPD SHARING:
Plan to Share IPD: Yes
Pfizer will provide access to individual de-identified participant data and related study documents (e.g. protocol, Statistical Analysis Plan (SAP), Clinical Study Report (CSR)) upon request from qualified researchers, and subject to certain criteria, conditions, and exceptions. Further details on Pfizer's data sharing criteria and process for requesting access can be found at: https://www.pfizer.com/science/clinical_trials/trial_data_and_results/data_requests.
URL: https://www.pfizer.com/science/clinical_trials/trial_data_and_results/data_requests

REFERENCES:
- See also: To obtain contact information for a study center near you, click here. — https://pmiform.com/clinical-trial-info-request?StudyID=B1851214

RESULTS

PARTICIPANT FLOW:
Recruitment Details: This study was conducted in India. Participants took part in the study for approximately 1 month.
Pre-assignment Details: A total of 200 participants were enrolled and vaccinated, all participants completed the 1-month follow-up after vaccination.
Groups:
- 13vPnC: Participants received 1 intramuscular dose of 13-valent pneumococcal conjugate vaccine (13vPnC) on Day 1.
Period: Vaccination Period
Arm/Group | 13vPnC
Started | 200
Completed | 200
Not Completed | 0
Period: 1-Month Follow-Up Period
Arm/Group | 13vPnC
Started | 200
Completed | 200
Not Completed | 0

BASELINE CHARACTERISTICS:
Population: All participants who received any study intervention and had safety data assessed after vaccination.
Arm/Group | 13vPnC
Number analyzed (Participants) | 200
Age, Continuous [Mean (Standard Deviation); unit: Years] | 31.4 (7.98)
Age, Continuous [Median (Full Range); unit: Years] | 29.0 [18 to 49]
Sex: Female, Male [Count of Participants; unit: Participants]
  Female | 92
  Male | 108
Race/Ethnicity, Customized [Count of Participants; unit: Participants]
  Race_Asian | 200
  Ethnicity_Non-Hispanic/Non-Latino | 200

OUTCOME MEASURES:

1. Primary Outcome: Percentage of Participants With Prompted Local Reactions Within 7 Days After Vaccination
Description: From Day 1 through Day 7 following vaccination, where Day 1 is the day of vaccination, local reactions including redness, swelling, and pain at the injection site were assessed and recorded.
Time Frame: Within 7 Days After Vaccination
Population: The safety population included all participants who received any study intervention and had safety data assessed after vaccination.
Measure: Number (95% Confidence Interval); unit: Percentage
Arm/Group | 13vPnC
Number analyzed (Participants) | 200
Percentage
  Redness | 1.5 [0.3 to 4.3]
  Swelling | 6.5 [3.5 to 10.9]
  Pain at Injection Site | 63.0 [55.9 to 69.7]

2. Primary Outcome: Percentage of Participants With Prompted Systemic Events Within 7 Days After Vaccination
Description: From Day 1 through Day 7 following vaccination, where Day 1 is the day of vaccination, systemic events including fever, headache, fatigue, muscle pain, and joint pain were assessed and recorded. Fever was defined as temperature ≥38.0 °C.
Time Frame: Within 7 Days After Vaccination
Population: as for outcome 1
Measure: Number (95% Confidence Interval); unit: Percentage
Arm/Group | 13vPnC
Number analyzed (Participants) | 200
Percentage
  Fever | 3.0 [1.1 to 6.4]
  Fatigue | 25.0 [19.2 to 31.6]
  Headache | 23.0 [17.4 to 29.5]
  Joint Pain | 7.5 [4.3 to 12.1]
  Muscle Pain | 32.0 [25.6 to 38.9]

3. Primary Outcome: Percentage of Participants With Adverse Events (AEs) Within 1 Month After Vaccination
Description: An AE was any untoward medical occurrence in a patient or clinical study participant, temporally associated with the use of study intervention, whether or not considered related to the study intervention. Local reactions (redness, swelling, and pain at the injection site) and systemic events (fever, headache, fatigue, muscle pain, and joint pain) were not collected as AEs.
Time Frame: Within 1 Month After Vaccination
Population: as for outcome 1
Measure: Number (95% Confidence Interval); unit: Percentage
Arm/Group | 13vPnC
Number analyzed (Participants) | 200
Percentage | 0.5 [0.0 to 2.8]

4. Primary Outcome: Percentage of Participants With Serious Adverse Events (SAEs) Within 1 Month After Vaccination
Description: An SAE was any untoward medical occurrence at any dose that resulted in death, was life-threatening (immediate risk of death), required inpatient hospitalization or prolongation of existing hospitalization, resulted in persistent or significant disability/incapacity (substantial disruption of the ability to conduct normal life functions), resulted in congenital anomaly/birth defect or considered to be an important medical event.
Time Frame: Within 1 Month After Vaccination
Population: as for outcome 1
Measure: Number (95% Confidence Interval); unit: Percentage
Arm/Group | 13vPnC
Number analyzed (Participants) | 200
Percentage | 0 [0 to 1.8]

ADVERSE EVENTS:
Time Frame: Within 1 month after vaccination.
Description: The same event may appear as both an AE and an SAE. However, what is presented are distinct events. An event may be categorized as serious in one participant and as non-serious in another participant, or one participant may have experienced both a serious and non-serious event during the study. The safety population were participants who received study intervention and had safety data assessed after vaccination.
Arm/Group | 13vPnC
All-Cause Mortality (participants affected / at risk) | 0/200
Serious Adverse Events (participants affected / at risk) | 0/200
Other Adverse Events (participants affected / at risk) | 1/200
OTHER ADVERSE EVENTS; cells are participants affected of the arm's N at risk (number of events):
Term (organ system) | 13vPnC (N=200)
Varicella (Infections and infestations) | 1 (1)

CERTAIN AGREEMENTS:
Principal investigators are sponsor employees: No; Agreement restricts PI disclosure of results: Yes; Restriction type: Other
Pfizer has the right to review disclosures, requesting a delay of less than 60 days. Investigator will postpone single center publications until after disclosure of pooled data (all sites), less than 12 months from study completion/termination at all participating sites. Investigator may not disclose previously undisclosed confidential information other than study results.

DOCUMENTS (2):
  • Study Protocol (2021-10-15): https://cdn.clinicaltrials.gov/large-docs/59/NCT05329259/Prot_000.pdf
  • Statistical Analysis Plan (2022-04-08): https://cdn.clinicaltrials.gov/large-docs/59/NCT05329259/SAP_001.pdf